CLINICAL TRIAL: NCT01948362
Title: A Randomised, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of Sulforadex® in Healthy Male Subjects
Brief Title: Sulforadex in Healthy Volunteers SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evgen Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVG001N
Record Dates: First submitted 2013-09-11; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Stage, Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — alpha-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulforadex (Active Comparator): Active compound
  Interventions: Drug: Sulforadex
- alpha Cyclodextrin (Experimental): Placebo control arm
  Interventions: Drug: Alpha cyclodextrin

INTERVENTIONS:
Drug: Sulforadex — Active compound
  Other Names: Stabilised sulforaphane
  Arms: Sulforadex
Drug: Alpha cyclodextrin — Placebo control
  Arms: alpha Cyclodextrin

SUMMARY:
To determine the safety and tolerability of single escalating doses of Sulforadex® in healthy male volunteers.

DETAILED DESCRIPTION:
This study will be conducted in a randomised, double-blind, placebo-controlled design with single ascending doses of Sulforadex® administered to healthy male subjects between 18 to 45 years of age. Each healthy subject will receive verbal and written information followed by signing of the Informed Consent Form (ICF).

Subjects will be screened within 21 days prior to admission. At this visit a medical examination will be performed to assess eligibility of the healthy subject. Screening will be conducted over 1 day or may be divided into more than 1 day. The first cohort of the study will commence with one sentinel group. The subsequent groups may be dosed together without sentinel dosing. The study is expected to have 5 cohorts with a total of 29 healthy male subjects:

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged between 18 and 45 years (inclusive) at screening.
2. Had a Body Mass Index (BMI) between 18.5 and 25.0 kg/m2 (inclusive) at screening.
3. Subjects agreed to use acceptable methods of contraception

Exclusion Criteria:

1. Subjects could not refrain from eating brassica vegetables or using brassica containing supplements for at least 7 days prior to the drug administration.
2. History or clinical evidence of clinically significant disease or any condition or disease that affects drug absorption, distribution or excretion.
3. Any history of clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission.
4. Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening and Day -1) and 24-hour 5-lead Holter ECG (at screening) which in the opinion of the Investigator interfered with the ECG analysis.
5. Any history or current evidence of clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological or psychiatric disease.
6. Positive screen for Hepatitis B (Hepatitis B surface Antigen, HBsAG), Hepatitis C (Hepatitis C Antibody, anti-HCV) or HIV.
7. Confirmed positive results from urine drug screen at screening and on admission (Day

   -1) indicating drug abuse including: amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, tricyclic antidepressants and methadone or a confirmed positive alcohol breath test at screening and on admission (Day -1).
8. History or clinical evidence of alcoholism or drug abuse. Alcohol abuse is defined as regular weekly intake of more than 14 units if female and 21 units if male (Using alcohol tracker http://www.nhs.uk/Tools/Pages/NHSAlcoholtracker.aspx); drug abuse is defined as compulsive, repetitive and/or chronic use of drugs or other substances with or without problems related to their use and/or where stopping or a reduction in dose will lead to withdrawal symptoms.
9. Subject was mentally handicapped.
10. Participation in another drug trial within 90 days prior to first drug administration.
11. Use of any medication (including over-the-counter [OTC] medication) within 2 weeks prior to admission (Day 1) or within 10 times the elimination half-life of the respective drug or anticipated concomitant medication during the treatment periods. Limited amounts of paracetamol were allowed to treat AEs.
12. Subjects who had donated more than 500 mL of blood within 90 days prior to drug administration.
13. Smoking more than 10 cigarettes or equivalent amount of tobacco per day and subjects who could not stop smoking for the duration of the study whilst in the CPU.
14. Treatment with herbal or sulforaphane containing supplements during the 7 days prior to dosing, or use of vitamins during 48 hours prior to admission (Day -1).
15. Any circumstances or condition(s) that in the opinion of the Investigator would compromise full participation in the trial or compliance with the protocol.
16. Subjects with legal incapacity or limited legal capacity at screening.
17. Subjects who were vegetarians, vegans or have medical dietary restrictions.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety | 2 days
  Safety assessments will include standard laboratory safety tests (haematology, biochemistry, coagulation and urinalysis), vital signs, physical examinations, 12-lead ECG, telemetry and AE monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Täube, MD FFPM, Principal Investigator — Richmond Pharmacology
Locations (1):
- Richmond Pharmacology, London, United Kingdom